CLINICAL TRIAL: NCT03851744
Title: The Mechanistic Effects of Acute Hypobaric Hypoxia on Exogenous Carbohydrate Utilization During Steady-state Aerobic Exercise
Brief Title: High Altitude and Exogenous Carbohydrate Oxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18-09HC
Record Dates: First submitted 2018-08-30; First posted 2019-02-22 (Actual); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Glucose Metabolism; High Altitude
MeSH Terms: conditions — Altitude Sickness | interventions — Sea Level Rise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sea Level (Active Comparator): Carbohydrate metabolism measured at SL
  Interventions: Other: Sea Level
- High Altitude (Experimental): Carbohydrate metabolism measured at HA
  Interventions: Other: High Altitude

INTERVENTIONS:
Other: Sea Level — Carbohydrate consumed at 1.8 g/min during treadmill exercise at SL
  Arms: Sea Level
Other: High Altitude — Carbohydrate consumed at 1.8 g/min during treadmill exercise at HA
  Arms: High Altitude

SUMMARY:
Recent studies have reported that oxidation of exogenous carbohydrate is reduced under acute hypobaric hypoxic (high altitude; HA) conditions compared to normoxia (sea level; SL) in native lowlanders. However, the mechanisms by which HA suppresses exogenous carbohydrate oxidation are not known. This study will seek to confirm that acute HA exposure decreases exogenous carbohydrate oxidation during steady-state aerobic exercise compared to SL, and explore if the mechanism inhibiting plasma glucose uptake is insulin dependent or independent.

DETAILED DESCRIPTION:
This randomized crossover study will examine substrate metabolic responses to ingesting supplemental carbohydrate during steady-state aerobic-type exercise at sea level (SL) and following acute (~5 h) exposure to HA (4,300 m) conditions in 10 healthy, recreationally active adults between the ages of 18-39 yrs. Following a 48-hr muscle glycogen normalization period, volunteers will complete 80-min of metabolically-matched, steady-state aerobic exercise on a treadmill, and consume 145 g of glucose (1.8 g·min-1) at SL and HA. Treadmill exercise will be performed at the same absolute workload, with speed and grade being the same at SL and HA to induce the same absolute workload between phases. SL and HA trials will occur in the US Army Research Institute of Environmental Medicine (USARIEM) hypobaric chamber and will be separated by a minimum 7-d washout period between each protocol day. 6-6-[2H2] glucose will be used as a tracer to assess glucose turnover. Indirect calorimetry, breath sampling for 13C/12C expired in CO2, and urine collections will be used to determine carbohydrate, fat, and protein oxidation during exercise at SL and HA. Serial blood draws will be collected during each trial to assess endocrine and circulating substrate responses to exercise, carbohydrate, and hypoxia. Muscle biopsies will be collected before and after steady-state exercise to examine intramuscular glucose transport expression and translocation, glycogen status, and activity enzyme intermediates in aerobic and anaerobic energy metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 - 39 years
* Born at altitudes less than 2,100 m (~7,000 feet; Examples include Santa Fe, New Mexico; Laramie, Wyoming; Etc.)
* Physically active based on assessment of physical activity history (2-4 days per week aerobic and/or resistance exercise)
* Have supervisor approval (permanent party military and civilians)
* Willing to refrain from alcohol, smokeless nicotine products and dietary supplement use during study periods
* Refrain from taking any nonsteroidal anti-inflammatory drugs (NSAIDs; e.g. aspirin, Advil®, Aleve®, Naprosyn®, or any aspirin-containing product) for 10 days before and at least 5 days AFTER each muscle biopsy. (*Tylenol® or acetaminophen is ok to use if needed for discomfort)

Exclusion Criteria:

* Born at altitudes greater than 2,100 m (~7,000 feet; Examples include Santa Fe, New Mexico; Laramie, Wyoming; Etc.)
* Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas that are more than 1,200 m for five days or more within the last 2 months (Examples include Ft. Huachuca, Arizona; Lima, Peru; Feldberg, Germany, Etc.)
* Musculoskeletal injuries that compromise exercise capability
* Metabolic or cardiovascular abnormalities (determined by resting ECG), gastrointestinal disorders (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Medication that affects macronutrient metabolism (i.e., diabetes medications, statins, corticosteroids, etc) and/or the ability to participate in strenuous exercise
* Evidence of apnea or other sleeping disorders
* Prior diagnosis of high altitude pulmonary edema (HAPE) or high altitude cerebral edema (HACE)
* Presence of asthma or respiratory tract infections (< 1 month prior)
* Allergies or intolerance to foods (including but not limited to lactose intolerance/milk allergy), vegetarian practices, or medications (including, but not limited to, lidocaine ) to be utilized in the study
* Smoking or vaping
* History of complications with lidocaine
* Taking medications that interfere with oxygen delivery and transport (Includes sedatives, sleeping aids, tranquilizers and/or any medication that depresses ventilation, diuretics, alpha and beta blockers)
* Evidence of any physical, mental, and/or medical conditions that would make the proposed studies relatively more hazardous as determined by the Office of Medical Support and Oversight
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Anemia (hematocrit <38% and hemoglobin <12.5 g/dL) and Sickle Cell Anemia/Trait
* Abnormal prothrombin time (PT)/ partial thromboplastin time (PTT) test or problems with blood clotting
* Blood donation within 8 weeks of beginning the study

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Margolis, PhD, Principal Investigator — Military Nutrition Division, USARIEM
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events happen prior to assignment of participants to a study arm.
Groups:
- Sea Level First, Then High Altitude: Carbohydrate metabolism measured at SL first then HA
  Sea Level: Carbohydrate consumed at 1.8 g/min during treadmill exercise at SL
  7 day washout
  High Altitude: Carbohydrate consumed at 1.8 g/min during treadmill exercise at HA
- High Altitude First, Then Sea Level: Carbohydrate metabolism measured at HA first then SL
  High Altitude: Carbohydrate consumed at 1.8 g/min during treadmill exercise at HA
  7 day washout
  Sea Level: Carbohydrate consumed at 1.8 g/min during treadmill exercise at SL
Period: Overall Study
Arm/Group | Sea Level First, Then High Altitude | High Altitude First, Then Sea Level
Started | 4 | 6
Completed | 4 | 4
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sea Level First, Then High Altitude: Carbohydrate metabolism measured at SL, then HA
  Sea Level: Carbohydrate consumed at 1.8 g/min during treadmill exercise at SL
  7 day washout
  High Altitude: Carbohydrate consumed at 1.8 g/min during treadmill exercise at HA
- High Altitude, Then Sea Level: Carbohydrate metabolism measured at HA, then SL
  High Altitude: Carbohydrate consumed at 1.8 g/min during treadmill exercise at HA
  7 day washout
  Sea Level: Carbohydrate consumed at 1.8 g/min during treadmill exercise at SL
- Total: Total of all reporting groups
Arm/Group | Sea Level First, Then High Altitude | High Altitude, Then Sea Level | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Rate of Exogenous Carbohydrate Oxidation
Description: Use indirect calorimetry and stable isotope methodologies to measure if acute HA exposure changes the rate of exogenous carbohydrate oxidation during steady-state aerobic exercise compared to SL
Time Frame: 7 hours
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | Sea Level | High Altitude
Number analyzed (Participants) | 8 | 8
g/min | 0.44 (0.05) | 0.35 (0.07)

2. Primary Outcome: Rate of Glucose Turnover
Description: Use stable isotope methodologies to measure if acute HA exposure changes the rate of glucose turnover during steady-state aerobic exercise compared to SL
Time Frame: 7 hours
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Sea Level | High Altitude
Number analyzed (Participants) | 8 | 8
mg/kg/min
  Glucose Rate of Disappearance | 14.3 (2.0) | 12.7 (1.7)
  Metabolic Clearance Rate | 12.1 (2.3) | 8.9 (1.8)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Sea Level | High Altitude
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03851744/Prot_SAP_000.pdf